CLINICAL TRIAL: NCT02332941
Title: Intravitreal Rituximab
Brief Title: Treatment -Resistant Neovascular Age-Related Macular Degeneration
Acronym: Rituximab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Rithwick Rajagopal, Assistant Professor, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201406106
Record Dates: First submitted 2014-10-28; First posted 2015-01-07 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): This is a pilot study. It will be an interventional, prospective, observational, clinical study that seeks to evaluate the effect of intravitreal rituximab over a period of one month.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — The purpose of this study is to determine if treatment of Age Related Macular Degeneration (AMD) with a new medication,rituximab is effective.

SUMMARY:
The purpose of this study is to determine if treatment of Age Related Macular Degeneration (AMD) with a new medication,rituximab is effective. To address this issue, investigators propose a clinical trial in which patients with late stage disease, poor vision and who have failed treatment by conventional means will receive rituximab by direct injection into the affected eye and will be followed for improvement in the structure of their retina. Age Related Macular Degeneration (AMD) is a leading cause of vision loss in the elderly with routine care involving injections in the eye to improve and to prevent worsening of vision. However, some patients do not respond to the medications that we currently have and as such an alternative medication is needed. One potential medication is rituximab, which has been injected into the eye for primary eye cancer, and has been tolerated well and led to patient improvement. Investigators will obtain baseline eye tests then plan on injecting this medication in to the eye of our patients with late stage AMD, by first placing numbing drops into the eye, then injecting the medication directly into the eye using sterile techniques. Investigators will then follow the patient and repeat eye tests to monitor for improvements.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 40
* Patients who have a diagnosis of wet age-related macular degeneration
* Patients who have a central visual acuity ,20/200
* Patients who have been deemed "treatment-resistant" at the discreation of the treating physician

Exclusion Criteria:

* Patients with treatment failure for neovascular AMD
* Patients who have tried multiple anti-vegf medication without anatomical or objective improvement

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Central Macular Thickness | 2 years
  Primary measure will be Central Macular Thickness as recorded with Optical Coherence Tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Rithwick Rajagopal, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States